CLINICAL TRIAL: NCT00100659
Title: Pegylated Interferon +/- Ribavirin for Children With Hepatitis C
Brief Title: PEDS-C: Pegylated Interferon +/- Ribavirin for Children With Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 67767 (completed); U01DK067767 (NIH)
Record Dates: First submitted 2005-01-04; First posted 2005-01-05 (Estimated); Results first posted 2013-07-01 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-08

CONDITIONS: Chronic Hepatitis C
Keywords: pediatric; hepatitis; children; HCV; PEG; PEG-2a; peginterferon alfa-2a; Pegylated Interferon; RV; ribavirin; Pegasys; CHC; chronic hepatitis C; chronic hepatitis C virus; hepatitis c; pediatric hepatitis; pediatric HCV
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis; Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Pegylated interferon/ribavirin (Active Comparator): Pegasys - 180 mcg per 1.73 meter squared body surface area subcutaneously once weekly.
  Ribavirin - 15 mg per kg orally twice daily using 100-mg tablets.
  Interventions: Drug: Pegylated Interferon/ribavirin
- Pegylated interferon/placebo (Placebo Comparator): Placebo tablets were supplied in the same dosing regimen as ribavirin, using the same number of tablets that would be given if ribavirin were being administered (eg, 3 placebo tablets twice daily for a 40-kg child who would receive 3 100-mg RV tablets twice daily).
  Interventions: Drug: Pegylated Interferon/ribavirin

INTERVENTIONS:
Drug: Pegylated Interferon/ribavirin

SUMMARY:
The purpose of this study is to determine the safety and efficacy of peginterferon alfa-2a (PEG-2a) in combination with ribavirin (RV) and PEG-2a alone for the treatment of chronic hepatitis C virus (CHC) infection in children.

The purpose of this study is also to determine whether PEG-2a in combination with RV or PEG-2a alone will result in a longer response rate in children with CHC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who are 5-18 years of age at enrollment (not yet reached 18th birthday at screening).
* HCV viremia (by any test) present on 2 tests separated by at least 6 months.
* Chronic liver disease, as indicated by inflammation and/or fibrosis, consistent with chronic hepatitis C infection on a liver biopsy obtained within the past 24 months, as assessed by a qualified pathologist, not consistent with other known liver disease and not normal.
* Compensated liver disease (Child-Pugh Grade A clinical classification)
* Signed informed consent from parent/legal guardian and willingness of parent/legal guardian to abide by the requirements of the study.
* Hemoglobin values >11 g/dL for females; > 12 g/dL for males
* Normal thyroid stimulating hormone (TSH)
* Able to swallow a ribavirin/placebo tablet

Exclusion Criteria:

* Any prior treatment with Interferon or ribavirin (RV)
* Receipt of any investigational drug <6 weeks prior to the first dose of study drug
* Any systemic antiviral therapy <6 weeks prior to the first dose of study drug. Exception: patients who have taken or are expected to require acyclovir for herpetic lesions
* Positive test at screening for anti-HAV IgM Ab, HBsAg, anti-HBc IgM Ab, or anti-HIV Ab
* History or other evidence of a medical condition associated with chronic liver disease other than HCV (abnormal ceruloplasmin, alpha-1-antitrypsin, ANA>1:160, SMA>1:80, anti-LKM antibody > 60 units))
* History or other evidence of bleeding from esophageal varices
* Decompensated liver disease (e.g. conjugated bilirubin >1.5mg/dl, ascites, varices, Child-Pugh Grade B or C clinical classification)
* History of autoimmune or immunologically mediated disease (e.g. inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, clinical evidence of rheumatoid arthritis)
* Absolute neutrophil count <1500 cells/mm3 , hemoglobin <11 g/dL for females and <12 g/dL for males, white blood count>17.5 x 109/L, or platelet count <90,000/ mm3
* Serum creatinine level >1.5 times the upper limit of normal for age
* Major depression according to the American Psychiatric Association, or a history of severe psychiatric disorder, such as major psychoses, suicidal ideation and/or suicide attempt
* History or other evidence of chronic pulmonary or cardiac disease associated with functional limitation
* History of thyroid disease poorly controlled on prescribed medications. Patients with elevated thyroid stimulating hormone (TSH) concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease are excluded
* Poorly controlled diabetes as defined by glycosylated hemoglobin of > 8%
* History of solid organ or bone marrow transplantation
* Evidence of severe retinopathy
* Coagulopathy (international normalized ratio>1.5)
* Evidence of an active or suspected cancer or a history of malignancy where the risk of recurrence is >20% within 2 years.
* Hemoglobinopathy
* Hemophilia
* Severe retinopathy
* History of other evidence of severe illness or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* Sexually active females of child-bearing potential (defined as age 10 years and older) and sexually active men who are not practicing two forms of effective contraception during treatment and during the 6 months after treatment has been concluded
* Females who have a positive serum pregnancy test within 7 days of initiation of treatment or who are breast-feeding
* Males whose female partners are pregnant
* Active substance abuse
* A sibling and/or any other child living in the same household or sharing the same primary caregiver enrolled in the study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Actual)
Dates: Start 2004-12; Primary Completion 2008-08 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen B Schwarz, MD, Principal Investigator — Johns Hopkins University
Locations (11):
- United States (11):
  - University of California, San Francisco, San Francisco, California
  - The Children's Hospital, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Indiana University School of Medicine, James Whitcomb Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital and Regional Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Protocols, manuals, and data will be posted at the NIDDK Central Repository
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data were posted to the NIDDK Central Repository in March 2013.
Access Criteria: Data can be requested from the NIDDK Central Repository. A signed data use agreement is required.
URL: https://repository.niddk.nih.gov/studies/peds-c/?query=peds-c

REFERENCES:
- [Background] Murray KF, Rodrigue JR, Gonzalez-Peralta RP, Shepherd J, Barton BA, Robuck PR, Schwarz KB; PEDS-C Clinical Research Network. Design of the PEDS-C trial: pegylated interferon +/- ribavirin for children with chronic hepatitis C viral infection. Clin Trials. 2007;4(6):661-73. doi: 10.1177/1740774507085445. PMID 18042575
- [Result] Rodrigue JR, Balistreri W, Haber B, Jonas MM, Mohan P, Molleston JP, Murray KF, Narkewicz MR, Rosenthal P, Smith LJ, Lobritto SJ, Schwarz KB, Robuck PR, Barton B, Gonzalez-Peralta RP. Peginterferon with or without ribavirin has minimal effect on quality of life, behavioral/emotional, and cognitive outcomes in children. Hepatology. 2011 May;53(5):1468-75. doi: 10.1002/hep.24248. PMID 21351116
- [Result] Schwarz KB, Gonzalez-Peralta RP, Murray KF, Molleston JP, Haber BA, Jonas MM, Rosenthal P, Mohan P, Balistreri WF, Narkewicz MR, Smith L, Lobritto SJ, Rossi S, Valsamakis A, Goodman Z, Robuck PR, Barton BA; Peds-C Clinical Research Network. The combination of ribavirin and peginterferon is superior to peginterferon and placebo for children and adolescents with chronic hepatitis C. Gastroenterology. 2011 Feb;140(2):450-458.e1. doi: 10.1053/j.gastro.2010.10.047. Epub 2010 Oct 28. PMID 21036173
- [Result] Goodman ZD, Makhlouf HR, Liu L, Balistreri W, Gonzalez-Peralta RP, Haber B, Jonas MM, Mohan P, Molleston JP, Murray KF, Narkewicz MR, Rosenthal P, Smith LJ, Robuck PR, Schwarz KB. Pathology of chronic hepatitis C in children: liver biopsy findings in the Peds-C Trial. Hepatology. 2008 Mar;47(3):836-43. doi: 10.1002/hep.22094. PMID 18167062
- [Result] Narkewicz MR, Rosenthal P, Schwarz KB, Drack A, Margolis T, Repka MX; PEDS-C Study Group. Ophthalmologic complications in children with chronic hepatitis C treated with pegylated interferon. J Pediatr Gastroenterol Nutr. 2010 Aug;51(2):183-6. doi: 10.1097/MPG.0b013e3181b99cf0. PMID 20512062
- [Result] Delgado-Borrego A, Gonzalez-Peralta RP, Raza R, Negre B, Goodman ZD, Jonas MM, Chung RT, Ludwig DA; PEDS-C Clinical Research Network. Correlates of adiponectin in hepatitis C-infected children: the importance of body mass index. J Pediatr Gastroenterol Nutr. 2015 Feb;60(2):165-70. doi: 10.1097/MPG.0000000000000604. PMID 25313851
- [Result] Schwarz KB, Molleston JP, Jonas MM, Wen J, Murray KF, Rosenthal P, Gonzalez-Peralta RP, Lobritto SJ, Mogul D, Pavlovic V, Warne C, Wat C, Thompson B. Durability of Response in Children Treated With Pegylated Interferon alfa [corrected] 2a +/- Ribavirin for Chronic Hepatitis C. J Pediatr Gastroenterol Nutr. 2016 Jan;62(1):93-6. doi: 10.1097/MPG.0000000000000929. PMID 26284539
- [Derived] Molleston JP, Mellman W, Narkewicz MR, Balistreri WF, Gonzalez-Peralta RP, Jonas MM, Lobritto SJ, Mohan P, Murray KF, Njoku D, Rosenthal P, Barton BA, Talor MV, Cheng I, Schwarz KB, Haber BA; PEDS-C Clinical Research Network. Autoantibodies and autoimmune disease during treatment of children with chronic hepatitis C. J Pediatr Gastroenterol Nutr. 2013 Mar;56(3):304-10. doi: 10.1097/MPG.0b013e3182774cae. PMID 23439301
- [Derived] Jonas MM, Balistreri W, Gonzalez-Peralta RP, Haber B, Lobritto S, Mohan P, Molleston JP, Murray KF, Narkewicz MR, Rosenthal P, Schwarz KB, Barton BA, Shepherd JA, Mitchell PD, Duggan C. Pegylated interferon for chronic hepatitis C in children affects growth and body composition: results from the pediatric study of hepatitis C (PEDS-C) trial. Hepatology. 2012 Aug;56(2):523-31. doi: 10.1002/hep.25690. Epub 2012 Jul 6. PMID 22383118

RESULTS

PARTICIPANT FLOW:
Recruitment Details: December 2004 to May 2006 at 11 US medical centers
Pre-assignment Details: Failure to meet inclusion criteria
Groups:
- Pegylated Interferon/Placebo: Placebo tablets were supplied in the same dosing regimen as ribavirin (RV), using the same number of tablets that would be given if ribavirin were being administered (eg, 3 placebo tablets twice daily for a 40-kg child who would receive 3 100-mg RV tablets twice daily).
Period: Overall Study
Arm/Group | Pegylated Interferon/Ribavirin | Pegylated Interferon/Placebo
Started | 55 | 59
Completed | 52 | 57
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pegylated Interferon/Ribavirin | Pegylated Interferon/Placebo | Total
Number analyzed (Participants) | 55 | 59 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 55 | 59 | 114
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.7 (3.3) | 10.8 (3.6) | 10.75 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 51
  Male | 27 | 36 | 63
Region of Enrollment [Number; unit: participants]
  United States | 55 | 59 | 114

OUTCOME MEASURES:

1. Primary Outcome: Sustained Viral Response (SVR)
Description: SVR is defined as nondetectable hepatitis C virus ribonucleic acid (HCV RNA) in plasma
Time Frame: at least 24 weeks after stopping treatment.
Measure: Number; unit: participants
Groups:
- PEG/RV: Pegylated interferon/ribavirin
- PEG/Placebo: Pegylated interferon/placebo
Arm/Group | PEG/RV | PEG/Placebo
Number analyzed (Participants) | 55 | 57
participants | 29 | 12

2. Secondary Outcome: Adverse Events
Description: Influenza-like, headache, and gastrointestinal symptoms
Time Frame: At any time up to 72 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Pegylated Interferon/Ribavirin: Pegasys - 180 mcg per 1.73 meter squared body surface area subcutaneously once weekly.
  Ribavirin - 15 mg per kg orally twice daily using 100-mg tablets.
  Pegylated Interferon/ribavirin
- Pegylated Interferon/Placebo: Placebo tablets were supplied in the same dosing regimen as ribavirin, using the same number of tablets that would be given if ribavirin were being administered (eg, 3 placebo tablets twice daily for a 40-kg child who would receive 3 100-mg RV tablets twice daily).
  Pegylated Interferon/ribavirin
Arm/Group | Pegylated Interferon/Ribavirin | Pegylated Interferon/Placebo
Number analyzed (Participants) | 55 | 57
Participants
  Influenza-like symptoms | 50 | 50
  Headache | 34 | 30
  Gastrointestinal symptoms | 31 | 37

ADVERSE EVENTS:
Arm/Group | Pegylated Interferon/Ribavirin | Pegylated Interferon/Placebo
Serious Adverse Events (participants affected / at risk) | 2/55 | 1/59
Other Adverse Events (participants affected / at risk) | 51/55 | 52/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Interferon/Ribavirin (N=55) | Pegylated Interferon/Placebo (N=59)
Suicide gesture (Psychiatric disorders) | 1 (1) | 0 (0) — Hospitalization
New onset diabetes mellitus Type 1 (Endocrine disorders) | 1 (1) | 0 (0) — Hospitalization
Complications of a liver biopsy (Hepatobiliary disorders) | 0 (0) | 1 (1) — Hospitalization and cholecystectomy
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated Interferon/Ribavirin (N=55) | Pegylated Interferon/Placebo (N=59)
Flu-like symptoms (General disorders) | 50 | 50
Headache (General disorders) | 34 | 30
Gastrointestinal symptoms (Gastrointestinal disorders) | 31 | 37
Injection site reaction (General disorders) | 25 | 27
Joint and muscle aches (Musculoskeletal and connective tissue disorders) | 20 | 20
Irritability (General disorders) | 17 | 13
Fatigue (General disorders) | 15 | 15
Rash (Skin and subcutaneous tissue disorders) | 11 | 14
Itching (Skin and subcutaneous tissue disorders) | 8 | 9
Anorexia (General disorders) | 7 | 11
Trouble sleeping (General disorders) | 6 | 11
Depression (Psychiatric disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less